CLINICAL TRIAL: NCT04217434
Title: A Comparative Evaluation of Various Patient Centered Outcomes Following Gingival Depigmentation Using Diode LASER in Different Modes: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Various Patient Centered Outcomes Following Gingival Depigmentation Using Diode LASER in Different Modes: A Randomized Clinical Trial
Acronym: LASER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, Head of the Department, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_D012_91556
Record Dates: First submitted 2019-12-12; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative; Healing Surgical Wounds; Analgesia; Temperature Change, Body
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 300µm in continous contact mode (Experimental): Diode LASER (A.R.C Fox , Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline.LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes , 300 µm fibre length will be used in continuous contact mode at a power setting of 1.5 to 3 W. • Simultaneously, increase in temperature on site will be recorded using FLUKETM 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain. Post operative instructions will be given.
  Interventions: Procedure: 300 µm fibre length will be used in continuous mode
- Group 300µm in pulsed contact mode (Experimental): Diode LASER (A.R.C Fox, Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline].LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes, 300 µm fibre length will be used in pulsed contact mode at a power setting of 1.5 - 3 W. Simultaneously, increase in temperature on site will be recorded using FLUKETM 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain. Post operative instructions will be given.
  Interventions: Procedure: 300 µm fibre length will be used in pulsed contact mode
- Group 400µm in continous contact mode (Experimental): Diode LASER (A.R.C Fox , Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline.LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes , 400 µm fibre length will be used in continuous contact mode at a power setting of 1.5 - 3 W. • Simultaneously, increase in temperature on site will be recorded using FLUKETM 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain. Post operative instructions will be given.
  Interventions: Procedure: 400 µm fibre length will be used in continuous contact mode
- Group 400µm in pulsed contact mode (Experimental): Diode LASER (A.R.C Fox , Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline.LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes , 400 µm fibre length will be used in pulsed contact mode at a power setting of 1.5 t 3 W. • Simultaneously, increase in temperature on site will be recorded using FLUKETM 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain. Post operative instructions will be given.
  Interventions: Procedure: 400 µm fibre length will be used in pulsed contact mode

INTERVENTIONS:
Procedure: 400 µm fibre length will be used in continuous contact mode — Diode LASER (A.R.C Fox, Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline].
  LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes using 400 µm fibre length will be used in continuous contact mode at a power setting of 1.5 - 3W. Simultaneously, increase in temperature on site will be recorded using FLUKE 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain.Post operative instructions will be given.
  Arms: Group 400µm in continous contact mode
Procedure: 400 µm fibre length will be used in pulsed contact mode — Diode LASER (A.R.C Fox, Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline].
  LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes using 400µm fibre length will be used pulsed contact mode at a power setting of 1.5 - 3W. Simultaneously, increase in temperature on site will be recorded using FLUKE 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain.Post operative instructions will be given.
  Arms: Group 400µm in pulsed contact mode
Procedure: 300 µm fibre length will be used in continuous mode — Diode LASER (A.R.C Fox, Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline].
  LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes using 300 µm fibre length will be used continous contact mode at a power setting of 1.5 - 3W. Simultaneously, increase in temperature on site will be recorded using FLUKE 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain.Post operative instructions will be given.
  Arms: Group 300µm in continous contact mode
Procedure: 300 µm fibre length will be used in pulsed contact mode — Diode LASER (A.R.C Fox, Germany, UK) with wavelength of 810nm is selected for the procedure. Before applying the LASER, operating staff and the patient will wear special LASER protective eye glasses.
  Local infiltration is administered with Lignox®[ 2% lignocaine in 1:80000 adrenaline].
  LASER tip will be used in contact mode on pigmented gingiva in short light paint brush strokes using 300 µm fibre length will be used pulsed contact mode at a power setting of 1.5 - 3W. .Simultaneously, increase in temperature on site will be recorded using FLUKE 59 Mini (IR) infrared thermometer in non contact mode. Water spray will be used to keep the area moist. Same procedure will be repeated till no pigments remain.Post operative instructions will be given.
  Arms: Group 300µm in pulsed contact mode

SUMMARY:
Purpose of this study is to clinically evaluate and compare various patient centered outcomes using diode LASER in Continuous mode (CW) and Pulsed Mode (PM) using 300µm and 400µm fiber for depigmentation procedure.

DETAILED DESCRIPTION:
The colour of gingiva has a tremendous impact on the esthetics of the smile. Clinically gingival melanin hyperpigmentation is presented as 'black gum' which is common esthetic problem especially for those who have gummy smile. Currently the growing aesthetic concerns among the patients require the removal of hyper pigmented gingival areas to create an aesthetically-pleasant smile. The harmony of the smile is determined not only by the shape, position and colour of the teeth or lips as well as by the by the gingival tissues.Several attempts have been made for removal of gingival pigmentation by different techniques like scalpel, electrocautery, LASER etc. Each technique has its own advantages and disadvantages. In the present study an effort has been made to compare two different modes viz. Continuous mode and Pulsed mode of LASER in the treatment of depigmentation.Diode LASERs for dentistry operate in the near infrared region. The most commonly used wavelengths are 810, 940 and 980 nm , because these wavelengths are very well absorbed by pigmented tissues, haemoglobin and melanin.There are several different ways LASER light operates: Continuous wave (CW), Pulse wave mode (PM). The continuous wave diodes emit continuous LASER energy with a fixed power output for the entire duration. Pulse modulated diodes create a 'pulse' by cutting the beam or turning LASER on & off [1s] at regular intervals.

During the first years of diode LASER treatment in dentistry only CW mode was possible but application of 3-4 Watt in CW mode led to carbonization of the soft tissue.To approach better results in soft tissue treatment without much carbonization it was necessary to interrupt the CW mode. That was done by chopping the CW mode. Pulses down to several 100μs were released.LASER in Continuous wave mode is suggested in some studies to cause increase in surgical site temperature which may cause necrosis or jeopardize healing. Application of the LASER in Pulsed mode prevents overheating of surrounding tissues. This study aims to determine the comparative increase in the onsite temperature between the two modes.Decrease in post-operative pain is likely to reduce the consumption of Non-steroidal Anti-inflammatory Drugs (NSAID's). The study aims to quantify the need for NSAID's post-operatively in both Pulsed and continuous wave modes and also in 300µ and 400µ fibers.

The change in the diameter of the fibers used in LASER irradiation could bring about a change in the outcome of the procedure as small diameter fibers means high energy density, faster cutting and more heat whereas with larger diameter fibers more energy is needed to cover a broader area to work more quickly and less heat.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of melanin hyper pigmentation of the anterior labial gingival segment
2. Systemically healthy patients who desires correction of gingival pigmentation
3. Patients with healthy periodontium
4. Patients in age group of 18-45 years old

Exclusion Criteria:

1. Presence of uncontrolled systemic diseases example uncontrolled Diabetes, Hypertension etc.
2. Pregnant and lactating women
3. Gingival enlargement
4. Patients who are on Non-steroidal Anti-inflammatory Drugs (NSAID's) or who have taken antibiotics for last 6 months
5. Patients who are on drugs that could possibly affect gingival status like phenytoin
6. Patients who have undergone any form of oral surgery in last 6 months
7. Asthma patients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-03-21 (Estimated); Study Completion 2020-11-22 (Estimated)

PRIMARY OUTCOMES:
pain assessing | 1st day post operatively.
  visual analogue scale (VAS) method - a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcomes.
pain assessing | 3rd day post operatively.
  visual analogue scale (VAS) method - a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcomes.
pain assessing | 7th day post operatively.
  visual analogue scale (VAS) method - a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcomes.
pain assessing | 14th day post operatively.
  visual analogue scale (VAS) method - a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcomes.
pain assessing | 1 month post operatively.
  visual analogue scale (VAS) method - a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcomes.
Healing of gingiva | 1st day post operatively
  hick healing index- score ranges from 0 to 4, higher values indicate the worst outcomes.
Healing of gingiva | 3rd day post operatively
  hick healing index- score ranges from 0 to 4, higher values indicate the worst outcomes.
Healing of gingiva | 7th day post operatively
  hick healing index- score ranges from 0 to 4, higher values indicate the worst outcomes.
Healing of gingiva | 14th day post operatively
  hick healing index- score ranges from 0 to 4, higher values indicate the worst outcomes.
Healing of gingiva | 1 month post operatively
  hick healing index- score ranges from 0 to 4, higher values indicate the worst outcomes.
epithelial healing | 7th day post operatively
  3% of hydrogen peroxide is applied on the operated area. no bubble- complete epithelization, bubble formation- incomplete epithelization.
epithelial healing | 14th day post operatively
  3% of hydrogen peroxide is applied on the operated area. no bubble- complete epithelization, bubble formation- incomplete epithelization.
epithelial healing | 1 month post operatively
  3% of hydrogen peroxide is applied on the operated area. no bubble- complete epithelization, bubble formation- incomplete epithelization.
need of analgesics | 1st day post operatively
  on scale of 0-9, where higher variable represents more pain
need of analgesics | 2nd day post operatively
  on scale of 0-9, where higher variable represents more pain
need of analgesics | 3rd day post operatively
  on scale of 0-9, where higher variable represents more pain
rise in temperature | baseline
  FLUKETM 59 Mini (IR) infrared thermometer is used to measure temperature at surgical site, more rise in temperature indicate more carbanoization.

SECONDARY OUTCOMES:
ease of cutting | Baseline
  on scale on 1-3, more value represents better cutting.
duration of operation | intraoperative
  time duration taken for completing surgical procedure in minutes
presence/ absence of carbonization | Baseline
  on scale of 0-3, higher value indicates more carbonization

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hafsa Shereen, MDS, Principal Investigator — Rajiv Gandhi University of Health Sciences; Dr Kishore H C, MDS, Study Director — Rajiv Gandhi University of Health Sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No